CLINICAL TRIAL: NCT01677130
Title: Standardized Application of High Frequency Oscillatory Ventilation in the Acute Respiratory Distress Syndrome (ARDS)
Status: Completed | Type: Observational
Sponsor: Ling Liu (Other)
Responsible Party: Sponsor-Investigator, Ling Liu, Physician Zhongda Hospital, Southeast University, China
Organization: Southeast University, China (Other)
Other Study IDs: FOV application
Record Dates: First submitted 2012-08-29; First posted 2012-08-31 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Clinical efficacy; safety; of HFOV treatment; of patients
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The Acute Respiratory Distress Syndrome (ARDS) is a clinical syndrome of progressive dyspnea and refractory hypoxemia caused by various reasons. Although in recent years a variety of supportive care measures have significant progress, but the mortality rate of patients with ARDS is still as high as 35-40%. Mechanical ventilation is one of the main treatments with ARDS, which is widely used in clinical. The rational mechanical ventilation strategy can improve the oxygenation of patients with ARDS and reduce lung injury. Patients with ARDS usually have alveolar epithelial and pulmonary capillary endothelial injury, and the lesion has heterogeneity. The protective mechanical ventilation strategies chosen by patients with ARDS in clinical practice are gradually being accepted and applied. The High-frequency oscillatory ventilation (HFOV) is a ventilation way with high respiratory rate and low tidal volume. Compared with conventional mechanical ventilation, HFOV may be able to more effectively improve oxygenation and reduce ventilator-associated lung injury. HFOV and protective ventilation strategy in ARDS is consistent with an important position in the treatment of ARDS, but not been widely adopted in clinical practice and is still only as a salvage treatment. Therefore, this study intends to use HFOV treatment with conventional mechanical ventilation by matching the cases in patients with ARDS. By comparing the influences of the patient's condition and mortality with HFOV, the clinical efficacy, safety, and health economics effectiveness of HFOV are further investigated and adaption time and parameter settings of HFOV are explored, which provide better treatment options for patients with ARDS and improve their prognosis.

ELIGIBILITY:
Inclusion Criteria:

* age> 18 years;
* lung protective ventilation (tidal volume 4-6ml/kg), airway plateau pressure is still higher than 30cmH2O, or the failure of conventional mechanical ventilation pneumothorax, bronchopleural fistula in patients with ARDS; of ARDS diagnosis in line with the 2012 Berlin ARDS diagnostic criteria.
* be able to sign informed consent.

Exclusion Criteria:

* severe pulmonary hemorrhage;
* severe intracranial high pressure;
* large airway stenosis and airway obstruction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients of ARDS age> 18 years
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2012-01; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)